CLINICAL TRIAL: NCT02711072
Title: Comparaison of Continuous Infusion of Local Anesthetic and Intrathecal Morphine for Pain Management in Elective Caeserean Section
Brief Title: Continuous Infusion for Pain Relief
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tunisian Military Hospital (Other)
Responsible Party: Principal Investigator, Dr trabelsi walid, associate professor, MD, Tunisian Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tunisian hh2
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Regional Anesthesia; Caeserian Section; Local Anesthetic
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Placebo Comparator)
  Interventions: Drug: control group; Drug: infiltration group
- infiltration group (Active Comparator)
  Interventions: Drug: control group; Drug: infiltration group

INTERVENTIONS:
Drug: control group — spinal anesthesia with 10 mg hyperbaric Bupivacaïne 0,5% + 2,5 µ Sufentanyl + 100 µ of intrathecal Morphine+ infiltration catheter with saline 5 ml/h
Drug: infiltration group — spinal anesthesia with 10 mg hyperbaric Bupivacaïne 0,5% + 2,5 µ Sufentanyl + 1ml of saline + infiltration catheter with 5 ml/h of Bupivacaïne 0,125%.

SUMMARY:
SPINAL anesthesia is commonly used for cesarean section, and it has become a popular practice to add opioids to spinal solutions to enhance and prolong intraoperative and postoperative analgesia. high incidence of side effects was noted. is there any alternative?

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* 18-45 years of age, inclusive
* elective caeserean section under spinal anesthesia

Exclusion Criteria:

* - contraindications to spinal anesthesia (e.g., allergy to local anesthetics, coagulopathy, malignancy or infection in the area)
* existing neurological deficit
* inability to understand the informed consent and demands of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analogic Scale | until 48 hours postoperative
  quality of postoperative analgesia

SECONDARY OUTCOMES:
occurrence of complications | 48 hours post operative
total dose of morphine consumption in mg | during 48 hours post operative

IPD SHARING:
Plan to Share IPD: Undecided